CLINICAL TRIAL: NCT03423238
Title: Targeting Obesity to Optimize Health in Cardiac Rehab (TOPCARE)
Acronym: TOPCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00046110; 1R56HL134989-01A1 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-06 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-09

CONDITIONS: Obesity; Weight Loss; CHD - Coronary Heart Disease
Keywords: Cardiac; Rehab; Diet; Exercise; Obese
MeSH Terms: conditions — Obesity; Weight Loss; Coronary Artery Disease; Motor Activity | interventions — Exercise; Caloric Restriction; Behavior Therapy; Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All assessments will take place by study staff blinded to the participant's treatment assignment. To ensure that staff remain blinded, participants will be asked not to discuss their intervention with the assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehab Only (Active Comparator): Patients will be randomized to Rehab only using a randomization scheme with blocking stratified by sex and obesity severity (BMI<30 vs. BMI≥30 kg/m2). All participants will undergo standard exercise-based cardiac rehabilitation, which includes meeting with dietitian, exercise, health education, and exercise compliance.
  Interventions: Other: Exercise; Behavioral: Health Education; Other: Exercise Compliance; Other: Dietary Counseling
- Rehab+Weight Loss (WL) (Experimental): Patients will be randomized to Rehab+WL using a randomization scheme with blocking stratified by sex and obesity severity (BMI<30 vs. BMI≥30 kg/m2). All participants will undergo standard exercise-based cardiac rehabilitation in addition to a weight-loss intervention, which includes meeting with dietitian, exercise, health education, and exercise compliance, calorie-restricted diet, behavioral modification, and weight-loss compliance.
  Interventions: Other: Exercise; Behavioral: Health Education; Other: Exercise Compliance; Dietary Supplement: Calorie-Restricted Diet; Behavioral: Behavioral Modification; Other: Weight-Loss Compliance

INTERVENTIONS:
Other: Exercise — Each exercise session lasts for 60 to 90 minutes and consists of 5-10 minutes of warm-up and cool-down activity; up to 30 minutes of aerobic exercise using a variety of modalities (e.g., walking laps on a track, cycle ergometry, treadmills, stair climbers); and 15-20 minutes of upper and lower body resistance exercises using Thera-Bands. An exercise physiologist creates an individualized plan
Behavioral: Health Education — Group education classes conducted by an exercise physiologist and/or dietitian are designed to provide support and general information on healthy lifestyle behaviors. Topics include risk factor control, diabetes, hypertension, lipids, medications, aerobic exercise, strength training and flexibility, weight control, reading food nutrition labels, eating out, holiday eating, intimacy, stress, relaxation, cardiac symptoms, and cardiac interventions.
Other: Exercise Compliance — Multiple behavioral management strategies to create a positive exercise environment and promote adherence and retention will be utilized. These include promptly contacting participants who miss a session, scheduling makeup sessions, and offering individual counseling sessions to discuss strategies to promote attendance and limit obstacles to participation.
Dietary Supplement: Calorie-Restricted Diet — Diet plans will provide a caloric deficit of 500 kcals per day. The lowest calorie level permitted will be 1,100 kcals for women and 1,200 kcals for men. The calorie distribution goal will be 15-20% from protein, <30% from fat, and 45-60% from carbohydrates. Participants will consume 2 meal replacements per day (Premier Protein shakes and bars); provided by the study)), along with one meal composed of traditional foods (500-750 kcals, low in fat, high in vegetables), and 1-3 snacks as needed (e.g., cereal bar, fruit, or vegetable, providing 100-150 kcals each). For the meal, patients will follow a weekly menu plan and recipes provided by the study. The food plan will be tailored to individual preferences and energy needs.
  Arms: Rehab+Weight Loss (WL)
Behavioral: Behavioral Modification — During months 1-3, participants will attend weekly individual behavioral counseling sessions with the study registered dietitian (RD); individual sessions will be held twice per month during months 4-6. The sessions will focus on self-monitoring, portion control, mindful eating, coping with negative thoughts, eating at regular times, and stress management. The RD will review individual progress, solve problems, answer questions, and set weight loss goals.
  Arms: Rehab+Weight Loss (WL)
Other: Weight-Loss Compliance — Participants will be asked to record their food and beverage intake in daily logs which will be reviewed weekly by the RD to verify compliance to the diet. Body weight will be measured weekly to ensure that participants are losing weight at an appropriate rate. If a participant is not meeting weight loss goals, energy intake will be modified accordingly to produce the desired rate of weight loss.
  Arms: Rehab+Weight Loss (WL)
Other: Dietary Counseling — Participants have one meeting with the Rehab dietitian upon starting.
  Arms: Rehab Only

SUMMARY:
Although coronary heart disease (CHD) treatment guidelines recognize obesity as a major modifiable risk factor,2 nearly half of all CHD patients are obese and the current standard of care fails to implement evidence-based obesity treatment for this high-risk population. Multiple lines of evidence suggest that weight loss improves outcomes in CHD patients. The primary goal of this study is to determine the feasibility of adding a 6-month behavioral weight loss intervention to exercise-based cardiac rehabilitation.

DETAILED DESCRIPTION:
Although coronary heart disease (CHD) treatment guidelines recognize obesity as a major modifiable risk factor,2 nearly half of all CHD patients are obese and the current standard of care fails to implement evidence-based obesity treatment for this high-risk population. The efficacy of exercise-based cardiac rehabilitation for improving exercise capacity and CHD risk factors is markedly blunted in CHD patients with obesity. Current programs largely focus on nutrient intake and produce minimal weight loss, on average. Our data show that despite appropriate exercise prescription and adherence, only 22% of CHD patients with obesity lose even the minimum recommended body weight over a 3-month program. These findings indicate that targeting reductions in caloric intake is needed to optimize outcomes in these patients and suggest that current programs are too short to produce adequate weight loss and ensure the necessary behavioral adaptations for long-term maintenance. Randomization to diet-induced weight loss in combination with aerobic exercise improves exercise capacity, quality of life, and CHD risk factors more than exercise alone and reduces long-term mortality in overweight and obese adults. The primary goal of this study is to determine the feasibility of adding a 6-month behavioral weight loss intervention to exercise-based cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* documented CHD defined as hospitalization for MI/heart attack coronary artery bypass grafting (CABG) or percutaneous coronary intervention (i.e., angioplasty, stent)
* age = 40 and older
* overweight or obese based on an elevated BMI (≥25 kg/m2)

Exclusion Criteria:

* body weight >450 lbs
* congestive heart failure (ejection fraction <35%)
* advanced kidney disease (on dialysis, or dialysis anticipated within 6 months)
* cognitive impairment (Montreal Cognitive Assessment [MoCA] score <22)
* major depression (Patient Health Questionnaire [PHQ-9] ≥20)
* severe pulmonary disease (i.e., oxygen-dependent)
* significant impairment from a prior stroke or other neurologic disease or injury
* high risk for non-adherence (i.e., unwilling or unable to comply with study requirements)
* current participation in physical therapy or another weight loss study
* current or recent use of weight loss medications (e.g., orlistat)
* prior weight loss procedure
* drug/substance abuse or excessive alcohol (> 14 drinks per week) within the past 6 months
* pregnant or pre-menopausal women
* peanut allergy
* milk allergy/lactose intolerance

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Brinkley, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Started | 19 | 19
Completed | 17 | 19
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rehab Only | Rehab+Weight Loss (WL) | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (7.9) | 63.5 (7.7) | 64.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 13 | 16 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 18 | 32
  Black | 3 | 1 | 4
  Hispanic | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Number of Enrolled Participants
Description: Total number of participants who met all inclusion/exclusion criteria and were enrolled in the study
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Includes all eligible participants prior to randomization
Arm/Group | All Participants
Number analyzed (Participants) | 38
Participants | 38

2. Primary Outcome: Compliance - Percentage of Sessions Attended
Description: The percentage of exercise/counseling sessions attended (calculated as the number of sessions attended divided by the number of sessions prescribed multiplied by 100)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of sessions attended
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 17 | 19
percentage of sessions attended
  Exercise compliance | 45.2 (27.5) | 68.6 (16.6)
  Dietary compliance | NA (NA) — Dietary compliance was not assessed in the Rehab Only group. | 98.2 (1.9)

3. Primary Outcome: Retention - Percentage of Participants Who Returned for Follow-up Testing
Description: The number of participants who returned for the 6-month follow-up visit divided by the total number of randomized participants multiplied by 100
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
Participants | 17 | 19

4. Secondary Outcome: Body Weight
Description: Body weight measured in kg
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
kg | 108.76 (19.32) | 102.85 (22.27)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.388, t-test, 2 sided

5. Secondary Outcome: Body Weight
Description: Body weight measured in kg
Time Frame: Months 3 and 6
Population: All available follow-up data were included. Rehab Only: 2 subjects dropped out prior to follow-up testing; 2 did not complete Month 3 testing due to a broken foot (n=1) and could not be reached (n=1); 5 did not complete Month 6 testing due to a COVID related pause on in-person research. Rehab+WL: 1 subject did not complete Month 6 testing due to a COVID related pause on in-person research.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 15 | 19
kg
  Month 3 | 104.852 (0.930) | 101.658 (0.854)
  Month 6: number analyzed (Participants) | 12 | 18
  Month 6 | 104.811 (1.290) | 99.122 (1.140)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.017, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.002, ANCOVA

6. Secondary Outcome: 6 Minute Walk (6MW) Test
Description: The 6MW test is a valid and reproducible measure of submaximal exercise capacity that reflects the level at which most activities of daily living are performed, predicts clinical events in cardiac patients, and is therefore a clinically meaningful outcome in cardiac rehabilitation studies. Participants were asked to walk at their own maximal pace on an established course, covering as much ground as they can during the allotted time, without running. Performance was measured by the total distance covered in meters.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
meters | 441.37 (81.86) | 429.47 (79.95)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.653, t-test, 2 sided

7. Secondary Outcome: 6 Minute Walk (6MW) Test
Description: as for outcome 6
Time Frame: Months 3 and 6
Population: All available follow-up data were included. Rehab Only: 2 subjects dropped out prior to follow-up testing; 3 did not complete Month 3 testing due to a broken foot (n=1), could not be reached (n=1), and safety/health concerns (n=1); 5 did not complete Month 6 testing due to a COVID related pause on in-person research. Rehab+WL: 1 subject did not complete Month 3 testing due to safety/health concerns; 1 did not complete Month 6 testing due to a COVID related pause on in-person research.
Measure: Geometric Least Squares Mean (Standard Error); unit: meters
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 14 | 18
meters
  Month 3 | 452.962 (10.935) | 446.916 (9.867)
  Month 6: number analyzed (Participants) | 12 | 18
  Month 6 | 448.506 (14.479) | 462.986 (12.668)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.684, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.458, ANCOVA

8. Secondary Outcome: Grip Strength
Description: Grip strength was measured twice in each hand using an isometric hydraulic hand dynamometer.
Time Frame: Baseline
Population: 2 participants (Rehab+WL) did not complete baseline testing due to safety/health concerns (n=2, Rehab+WL).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 17
kg | 34.21 (8.74) | 35.94 (8.40)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.550, t-test, 2 sided

9. Secondary Outcome: Grip Strength
Description: Grip strength was measured twice in each hand using an isometric hydraulic hand dynamometer.
Time Frame: Months 3 and 6
Population: All available follow-up data were included. Rehab Only: 2 subjects dropped out prior to follow-up testing; 2 did not complete Month 3 testing due to a broken foot (n=1) and could not be reached (n=1); 5 did not complete Month 6 testing due to a COVID related pause on in-person research. Rehab+WL: 2 subjects did not complete Month 3 testing due to safety/health concerns; 3 did not complete Month 6 testing due to a COVID related pause on in-person research (n=1) or safety/health concerns (n=2).
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 15 | 17
kg
  Month 3 | 33.711 (1.242) | 33.652 (1.182)
  Month 6: number analyzed (Participants) | 12 | 16
  Month 6 | 34.534 (1.218) | 35.837 (1.082)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.973, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.432, ANCOVA

10. Secondary Outcome: Mobility - MAT-sf
Description: Mobility was assessed using the MAT-sf, a 10-item computer-based, self-administered assessment that uses animated video clips of 10 different tasks to illustrate various mobility-related challenges that cover a broad range of functioning. Participants provide an assessment of their ability to perform each task on the computer by clicking the appropriate response (yes/no, number of minutes, number of times). Scores range from 30 to 80, with higher scores indicative of better mobility.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
score on a scale | 64.87 (8.72) | 61.47 (8.44)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.23063, t-test, 2 sided

11. Secondary Outcome: Mobility - MAT-sf
Description: as for outcome 10
Time Frame: Months 3 and 6
Population: All available follow-up data were included. Rehab Only: 2 subjects dropped out prior to follow-up testing; 3 did not complete Month 3 testing due to a broken foot (n=1), could not be reached (n=1), and technical difficulties (n=1); 5 did not complete Month 6 testing due to a COVID related pause on in-person research. Rehab+WL: 1 subject did not complete Month 6 testing due to a COVID related pause on in-person research.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 14 | 19
score on a scale
  Month 3 | 64.839 (1.484) | 65.212 (1.332)
  Month 6: number analyzed (Participants) | 12 | 18
  Month 6 | 64.613 (2.144) | 65.069 (1.848)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.854, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.874, ANCOVA

12. Secondary Outcome: Expanded Short Physical Performance Battery (eSPPB)
Description: The expanded Short Physical Performance Battery (eSPPB) is a modified version of a widely used assessment of lower extremity physical function that consists of 3 standing balance tasks held for 10 seconds each (side-by-side, tandem and semi-tandem), two 4-m walk tests to assess usual gait speed, and 5 repeated chair stands. To minimize ceiling effects and maximize overall dispersion of test scores, the eSPPB increases the holding time of the semi- and full-tandem stands to 30 seconds and adds a single leg stand and a narrow walk test of balance (walking at usual pace within lines of tape spaced 20 cm apart). eSPPB scores are continuous and range from 0 to 4, with higher scores indicative of better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
score on a scale | 1.99 (0.42) | 2.08 (0.55)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.563, t-test, 2 sided

13. Secondary Outcome: Expanded Short Physical Performance Battery (eSPPB)
Description: as for outcome 12
Time Frame: Months 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 15 | 19
score on a scale
  Month 3 | 2.252 (0.069) | 1.992 (0.061)
  Month 6: number analyzed (Participants) | 12 | 18
  Month 6 | 2.121 (0.110) | 2.135 (0.091)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.008, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.922, ANCOVA

14. Secondary Outcome: Health-related Quality of Life SF-36 - Mental Component Summary (MCS) Score
Description: Health-related quality of life was assessed using the Medical Outcomes Study Short Form 36 (SF-36), a 36-item self-report measure with well-documented psychometric properties across a wide range of populations. All items are scored on a 0 to 100 range such that a high score defines a more favorable quality of life. The SF-36 generates eight subscale scores (general health perceptions; physical functioning; role limitations due to physical problems; bodily pain; mental health; role limitations due to emotional problems; vitality; and social functioning) which are generated by averaging items in the same subscale. The mental component summary (MCS) score is derived using a factor analysis technique that includes positive weights for the vitality, social functioning, role-emotional, and mental health scales and negative weights for the physical functioning, role-physical, bodily pain and general health scales.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
score on a scale | 54.92 (8.52) | 53.50 (11.45)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.667, t-test, 2 sided

15. Secondary Outcome: Health-related Quality of Life SF-36 - Mental Component Summary (MCS) Score
Description: as for outcome 14
Time Frame: Months 3 and 6
Population: All available follow-up data were included. Rehab Only: 2 subjects dropped out prior to follow-up testing; 2 did not complete Month 3 testing due to a broken foot (n=1) and could not be reached (n=1).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 17 | 19
score on a scale
  Month 3: number analyzed (Participants) | 15 | 19
  Month 3 | 54.778 (2.003) | 53.698 (1.820)
  Month 6 | 53.885 (2.107) | 55.463 (1.995)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.692, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.590, ANCOVA

16. Secondary Outcome: Health-related Quality of Life SF-36 - Physical Component Summary (PCS) Score
Description: Health-related quality of life was assessed using the Medical Outcomes Study Short Form 36 (SF-36), a 36-item self-report measure with well-documented psychometric properties across a wide range of populations. All items are scored on a 0 to 100 range such that a high score defines a more favorable quality of life. The SF-36 generates eight subscale scores (general health perceptions; physical functioning; role limitations due to physical problems; bodily pain; mental health; role limitations due to emotional problems; vitality; and social functioning) which are generated by averaging items in the same subscale. The physical component summary (PCS) score is derived using a factor analysis technique that includes positive weights for the physical functioning, role-physical, bodily pain, general health and vitality scales and negative weights for the social functioning, role-emotional and mental health scales.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
score on a scale | 37.97 (10.51) | 37.30 (10.17)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.844, t-test, 2 sided

17. Secondary Outcome: Health-related Quality of Life SF-36 - Physical Component Summary (PCS) Score
Description: as for outcome 16
Time Frame: Months 3 and 6
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 17 | 19
score on a scale
  Month 3: number analyzed (Participants) | 15 | 19
  Month 3 | 42.458 (1.771) | 41.595 (1.615)
  Month 6 | 41.949 (2.374) | 42.569 (2.245)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.721, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.851, ANCOVA

18. Secondary Outcome: Arterial Stiffness
Description: Arterial stiffness was assessed as carotid-femoral pulse wave velocity (PWV). Carotid-femoral PWV was measured in the supine position using the SphygmoCor XCEL system. PWV is calculated by dividing the distance between the carotid and femoral arteries by the pulse transit time.
Time Frame: Baseline
Population: 15 participants (n=8, Rehab Only; n=7, Rehab+WL) did not complete baseline PWV testing due to technical difficulties (i.e., equipment malfunction, could not acquire signal); 1 participant (Rehab Only) refused.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 10 | 12
m/s | 8.67 (2.53) | 8.40 (2.73)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.815, t-test, 2 sided

19. Secondary Outcome: Arterial Stiffness
Description: as for outcome 18
Time Frame: Months 3 and 6
Population: All available follow-up data were included. Rehab Only: 2 subjects dropped out prior to follow-up testing; 8 did not complete Month 3 testing due to a broken foot (n=1), could not be reached (n=1), and technical issues (n=6); 11 did not complete Month 6 testing due to a COVID related pause (n=5) and technical issues (n=6). Rehab+WL: 2 subjects did not complete Month 3 testing due to technical issues; 4 did not complete Month 6 testing due to a COVID related pause (n=1) and technical issues (n=3)
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 9 | 17
m/s
  Month 3 | 8.760 (0.768) | 8.061 (0.616)
  Month 6: number analyzed (Participants) | 6 | 15
  Month 6 | 9.611 (0.719) | 8.487 (0.567)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.488, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.237, ANCOVA

20. Secondary Outcome: Brachial Blood Pressure - Systolic
Description: Brachial blood pressure was measured using a conventional mercury sphygmomanometer with the participant in a seated position after resting quietly for 5-10 minutes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
mmHg | 132.84 (21.14) | 128.63 (17.30)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Test type: Superiority; p = 0.506, t-test, 2 sided

21. Secondary Outcome: Brachial Blood Pressure - Systolic
Description: as for outcome 20
Time Frame: Months 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 15 | 19
mmHg
  Month 3 | 124.089 (3.564) | 126.987 (3.178)
  Month 6: number analyzed (Participants) | 12 | 18
  Month 6 | 124.272 (4.110) | 129.860 (3.399)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.549, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.303, ANCOVA

22. Secondary Outcome: Brachial Blood Pressure - Diastolic
Description: as for outcome 20
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
mmHg | 76.26 (14.02) | 75.89 (13.26)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.934, t-test, 2 sided

23. Secondary Outcome: Brachial Blood Pressure - Diastolic
Description: as for outcome 20
Time Frame: Months 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 15 | 19
mmHg
  Month 3 | 70.024 (2.166) | 69.247 (1.962)
  Month 6: number analyzed (Participants) | 12 | 18
  Month 6 | 72.738 (2.546) | 69.989 (2.168)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.792, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.417, ANCOVA

24. Secondary Outcome: Aortic Blood Pressure - Systolic
Description: Aortic blood pressure was measured using the SphygmoCor XCEL system with the participant in the supine position after resting quietly for 5-10 minutes.
Time Frame: Baseline
Population: 1 participant (Rehab Only) did not complete baseline testing due to safety/health concerns.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 18 | 19
mmHg | 132.89 (19.33) | 130.47 (16.57)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.685, t-test, 2 sided

25. Secondary Outcome: Aortic Blood Pressure - Systolic
Description: Aortic blood pressure was measured using the SphygmoCor XCEL system with the participant in a supine position after resting quietly for 5-10 minutes.
Time Frame: Months 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 15 | 19
mmHg
  Month 3 | 130.234 (3.650) | 129.328 (3.255)
  Month 6: number analyzed (Participants) | 12 | 18
  Month 6 | 127.204 (3.203) | 126.692 (2.647)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.854, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.903, ANCOVA

26. Secondary Outcome: Aortic Blood Pressure - Diastolic
Description: as for outcome 25
Time Frame: Baseline
Population: 1 participant (Rehab Only) did not complete baseline testing due to safety/health concerns.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 18 | 19
mmHg | 83.72 (15.23) | 81.11 (12.36)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.569, t-test, 2 sided

27. Secondary Outcome: Aortic Blood Pressure - Diastolic
Description: as for outcome 25
Time Frame: Months 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 15 | 19
mmHg
  Month 3 | 78.322 (2.127) | 78.965 (1.905)
  Month 6: number analyzed (Participants) | 12 | 18
  Month 6 | 76.221 (2.307) | 78.783 (1.924)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.824, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.401, ANCOVA

28. Secondary Outcome: Hemoglobin A1c
Description: Hemoglobin A1c was measured in whole blood using a turbidimetric inhibition immunoassay.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin glycated
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
percentage of hemoglobin glycated | 6.36 (0.97) | 5.94 (0.96)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.188, t-test, 2 sided

29. Secondary Outcome: Hemoglobin A1c
Description: Hemoglobin A1c was measured in whole blood using a turbidimetric inhibition immunoassay.
Time Frame: Months 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin glycated
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 15 | 19
percentage of hemoglobin glycated
  Month 3 | 6.046 (0.143) | 6.239 (0.134)
  Month 6: number analyzed (Participants) | 12 | 18
  Month 6 | 6.033 (0.163) | 6.190 (0.148)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.338, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.484, ANCOVA

30. Secondary Outcome: Fasting Insulin
Description: Insulin was determined by a chemiluminescent immunoassay.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 19 | 19
mg/dl | 22.67 (14.24) | 20.08 (10.89)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Baseline; Test type: Superiority; p = 0.533, t-test, 2 sided

31. Secondary Outcome: Fasting Insulin
Description: Insulin was determined by a chemiluminescent immunoassay.
Time Frame: Months 3 and 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
Number analyzed (Participants) | 15 | 19
mg/dl
  Month 3 | 20.161 (2.626) | 20.197 (2.414)
  Month 6: number analyzed (Participants) | 12 | 18
  Month 6 | 17.558 (3.276) | 19.623 (2.878)
Statistical Analysis 1: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 3; Test type: Superiority; p = 0.992, ANCOVA
Statistical Analysis 2: Comparison: Rehab Only vs Rehab+Weight Loss (WL); Month 6; Test type: Superiority; p = 0.639, ANCOVA

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Rehab Only | Rehab+Weight Loss (WL)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/19 | 0/19
Other Adverse Events (participants affected / at risk) | 10/19 | 10/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rehab Only (N=19) | Rehab+Weight Loss (WL) (N=19)
Angina/Percutaneous coronary intervention procedure (Cardiac disorders) | 1 (1) | 0 (0)
Left basilar pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rehab Only (N=19) | Rehab+Weight Loss (WL) (N=19)
acute bronchitis and URI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back Pain-Pinched nerve (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
bilateral feet and leg pain, left leg and foot pain worse (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
bilateral hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bleeding diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhea and Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
elevated BP and low oxygen/wound (Cardiac disorders) | 0 (0) | 1 (1)
Facial Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flu (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Flu symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Groin strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
left ankle fracture and left midfoot fractures (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
left hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
left knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
left leg injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nauseous possibly due to low blood sugar (Gastrointestinal disorders) | 0 (0) | 1 (1)
Outpatient ablation procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
pink eye (Eye disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postural Dizziness with presynscope (Cardiac disorders) | 1 (1) | 0 (0)
pre-planned outpatient ablation procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Pulled muscle in back and left knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
right ankle and heel pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sinus allergy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Strep Throat and flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fluid overload and increasing shortness of breath (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood loss (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT03423238/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT03423238/ICF_002.pdf